CLINICAL TRIAL: NCT00124397
Title: Effect of High Dose Statin Therapy on Endothelial Function in Patients With Type 2 Diabetes Mellitus Without CAD
Brief Title: Atorvastatin and Endothelial Function in Type 2 Diabetes Mellitus (ATTEND-Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20000084; 2162
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2005-08-05 (Estimated); Status verified 2005-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The aim of this study is to examine the effect of intensive cholesterol lowering therapy and tight blood pressure (BP) regulation on endothelial function (inner cell layer of vessels that determines dilatation) in type 2 diabetic patients without documented cardiovascular (CV) disease. The hypothesis is that intensive cholesterol lowering and tight blood pressure regulation will due better than a control group.

DETAILED DESCRIPTION:
Background:The prevalence of diagnosed type 2 diabetes mellitus (DM) is estimated to 2-4% in the general population in most European countries. DM is associated with an increased frequency of manifest atherosclerotic disease. Data from prospective studies demonstrate that the risk of developing acute coronary syndrome (ACS) in diabetic patients with no prior history of coronary artery disease (CAD) is equivalent to the risk observed in non-diabetics ACS survivors. Most diabetic patients die from CAD. Although DM is primarily a metabolic disorder, it imposes a tremendous burden on macro- and micro-vessel disease.The important question of primary prevention of cardiovascular disease (CVD) in DM remains unanswered.

In the major lipid-intervention studies where patients with CAD were included, the subgroup with DM had at least as good effect of lipid lowering therapy with statins as non-diabetics. The recently published Heart Protection Study supports the hypothesis of a favourable effect of statins in the primary prevention of CVD in DM. The UK Prospective Diabetic Study has proved that tight blood pressure (BP) regulation reduces the frequency of micro- and macrovascular endpoint. It has been suggested that combined lipid lowering with statins and tight BP regulation can have an additive effect in DM patients.

It is well established that the atherosclerotic process has an impact on endothelial function.An improvement of endothelial function by cholesterol lowering and BP reduction may serve as a surrogate endpoint for CAD.

Objective:To assess the effect of intensive lipid lowering on endothelial function in patients with DM and serum cholesterol level <6.5 mmol/l and to evaluate the effect of combined lipid lowering and tight BP regulation on endothelial function in the same patient group.

Methods: This is a single-center, randomised, placebo-controlled study with three treatment arms. Participants are blindly allocated to: 1. atorvastatin 80 mg daily 2. corresponding placebo 3. open label treatment with atorvastatin 80 mg daily and tight BP regulation with 5-10 mg amlodipine, 2-4 mg perindopril, 4-8 mg doxazosin in mono- or combination therapy that aims BP <130/80.

Endothelial function is evaluated at baseline, at 6 and 12 month non-invasively. A high resolution ultrasound scan is performed on the right brachial artery to assess post ischemic flow mediated changes in arterial diameter. Flow mediated dilatation (FMD) depends on an intact endothelium and is mediated via endogenous nitric oxid (NO). To test non-endothelium dependent vasodilatation 0.4 mg of sublingual nitroglycerin (NG) is administrated. NG is a smooth muscle relaxant and acts as a source of NO.There is a well described relation tween endothelial function in the coronary arteries and in the brachial artery.

Sample size: the sample size in the study is based on the following assumptions:

1. High resolution ultrasound technique has a high accuracy and reproducibility.
2. The majority of the patients will have endothelial dysfunction
3. As shown in previous clinical studies, an increase in FMD of 2% is significant at the 95% confidence interval.
4. Patients randomised to atorvastatin will after one year treatment show an improvement of FMD of at leat 2% compared with the placebo group. Patients treated openly with atorvastatin and BP regulation will have a further improvement of FMD of 2%.

Under these assumptions with a power of 80% and a 2 sided alfa of 5% a sample size of 160 patients are needed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus,
* Total cholesterol <6.5 mmol/l
* Signed informed consent

Exclusion Criteria:

* Documented CAD or peripheral vascular disease
* Treatment with lipid-lowering drugs
* Contraindications to HMG-CoA reductase therapy
* Potential noncompliance

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186
Dates: Start 2001-07; Study Completion 2004-12

PRIMARY OUTCOMES:
Flow mediated vasodilatation (FMD) on atorvastatin

SECONDARY OUTCOMES:
FMD on combined treatment
FMD in relation to lipid levels
FMD in relation to BP lowering
CV events

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, MD, Study Chair — Department of Medical Research, SHF Svendborg
Locations (1):
- Department of Medical Research, SHF Svendborg, Svendborg, Denmark